CLINICAL TRIAL: NCT06225596
Title: A Randomized Open-Label Phase 2/3 Study of BT8009 as Monotherapy or in Combination in Participants With Locally Advanced or Metastatic Urothelial Cancer (Duravelo-2)
Brief Title: Study BT8009-230 in Participants With Locally Advanced or Metastatic Urothelial Cancer (Duravelo-2)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BicycleTx Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT8009-230; 2023-504231-41 (EudraCT Number); U1111-1300-3791 (Other: UTN)
Record Dates: First submitted 2024-01-12; First posted 2024-01-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Urothelial Cancer
Keywords: Metastatic Urothelial Cancer; BT8009; Bladder cancer; Pembrolizumab; Chemotherapy; Avelumab; Zelenectide pevedotin
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; Gemcitabine; Cisplatin; Carboplatin; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: BT8009 Arm 1 (Experimental): Participants will receive BT8009 and a standard dose of pembrolizumab.
  Interventions: Drug: BT8009; Drug: Pembrolizumab
- Cohort 1: BT8009 Arm 2 (Experimental): Participants will receive BT8009 and a standard dose of pembrolizumab.
  Interventions: Drug: BT8009; Drug: Pembrolizumab
- Cohort 1: Arm 3 (Active Comparator): Participants will receive Platinum-based combination chemotherapy +/- avelumab maintenance
  Interventions: Drug: Gemcitabine + cisplatin Or carboplatin; Drug: Avelumab
- Cohort 2: BT8009 Arm 1 (Experimental): Participants will receive BT8009.
  Interventions: Drug: BT8009
- Cohort 2: BT8009 Arm 2 (Experimental): Participants will receive BT8009.
  Interventions: Drug: BT8009
- Cohort 2: Arm 3: BT8009 (Not Recruiting) (Experimental): Participants will receive BT8009 and a standard dose of pembrolizumab.
  Interventions: Drug: BT8009; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BT8009 — Participants will receive BT8009 on Days 1, 8, and 15 of every 21-day cycle.
  Arms: Cohort 1: BT8009 Arm 1; Cohort 2: BT8009 Arm 1
Drug: BT8009 — Participants will receive BT8009 on Days 1 and 8 of every 21-day cycle.
  Arms: Cohort 1: BT8009 Arm 2; Cohort 2: BT8009 Arm 2
Drug: BT8009 — Participants will receive BT8009 on days 1, 8 +/- 15 schedule of every 21-day cycle.
  Arms: Cohort 2: Arm 3: BT8009 (Not Recruiting)
Drug: Pembrolizumab — Participants will receive Pembrolizumab on Day 1 of every 21-day cycle. Pembrolizumab infusion will be started 30 minutes following the completion of the BT8009 infusion.
  Arms: Cohort 1: BT8009 Arm 1; Cohort 1: BT8009 Arm 2; Cohort 2: Arm 3: BT8009 (Not Recruiting)
Drug: Gemcitabine + cisplatin Or carboplatin — Participants will receive Gemcitabine on Days 1 and 8 of every 21-day cycle plus cisplatin Or carboplatin on Day 1 of every 21-day cycle.
  Arms: Cohort 1: Arm 3
Drug: Avelumab — After 4-6 cycles of Gemcitabine + Cisplatin or Carboplatin participants will receive maintenance Avelumab, if clinically indicated, on Days 1 and 15 each 28-day cycle.
  Arms: Cohort 1: Arm 3

SUMMARY:
This is a global, multicenter, randomized, open-label study, with an adaptive design. The main objective of the study is to measure the efficacy and safety of BT8009 (zelenectide pevedotin) as monotherapy and in combination with pembrolizumab in participants with locally advanced or metastatic urothelial cancer (UC). The study includes a dose selection phase followed by an adaptive design continuation. The study is comprised of 2 cohorts. Cohort 1 will include participants who have not received any prior systemic therapy for locally advanced or metastatic UC and are eligible to receive platinum-based chemotherapy, whereas Cohort 2 will include participants who have received ≥ 1 prior systemic therapy for locally advanced or metastatic UC.

ELIGIBILITY:
Key Inclusion Criteria:

* Life expectancy ≥ 12 weeks.
* Measurable disease as defined by RECIST v1.1.
* Histologically or cytologically confirmed locally advanced (unresectable) or metastatic UC of the renal pelvis, ureter, bladder, or urethra.
* Archival or fresh tumor tissue comprising muscle-invasive UC or locally advanced or metastatic UC should be available for submission to central laboratory.
* Negative pregnancy test for women of childbearing potential (WOCBP) (negative serum test at Screening and negative urine or serum test within 72 hours prior to the first dose).
* Cohort 1: Previously Untreated: Eligible to receive platinum-based chemotherapy (either cisplatin- or carboplatin-based chemotherapy based on Investigator decision.
* Cohort 1: Participants must not have received prior systemic therapy for locally advanced or metastatic UC with the following exceptions:

  1. Prior local intravesical chemotherapy, local surgery when full resection is not achieved, local immunotherapy, and radiotherapy are permitted if completed at least 4 weeks prior to the initiation of study treatment and all acute toxicities have resolved.
  2. Prior neoadjuvant/adjuvant chemotherapy or monomethyl auristatin E (MMAE)-based therapy with recurrence >12 months from completion of therapy.
  3. Prior neoadjuvant/adjuvant immune checkpoint inhibitor therapy with recurrence >12 months from completion of therapy.
* Cohort 2: Previously Treated: Participants must have received ≥ 1 prior systemic treatment for locally advanced or metastatic UC. This includes neoadjuvant/adjuvant platinum-based chemotherapy if recurrence occurred within 12 months of completing therapy.
* Cohort 2: Progression or recurrence of UC during or following receipt of most recent therapy.

Key Exclusion Criteria:

* Active keratitis or corneal ulcerations.
* Requirement, while on study, for treatment with strong inhibitors or strong inducers of human cytochrome P450 3A (CYP3A) or inhibitors of P-glycoprotein (P-gp) including herbal- or food-based inhibitors.
* Any condition requiring current treatment with high dose corticosteroids (> 10 mg daily prednisone or equivalent).
* Known hypersensitivity or allergy to any of the ingredients of any of the study interventions, or to MMAE.
* Has not adequately recovered from recent major surgery (excluding placement of vascular access).
* Receipt of live or attenuated vaccine within 30 days of first dose.
* Cohort 1: Previously Untreated: Prior treatment with a checkpoint inhibitor (CPI) for any other malignancy within the last 12 months.
* Cohort 2: Previously Treated: Received more than 1 prior platinum-based chemotherapy regimen for locally advanced or metastatic UC. This includes neoadjuvant/adjuvant platinum-based chemotherapy if recurrence occurred within 12 months of completing therapy.
* Cohort 2: Prior treatment with enfortumab vedotin or any other MMAE-based therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 956 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) assessed by blinded central independent review (BICR) | Up to approximately 6 years
  The time from randomization to date of first documentation of disease progression or death.
Cohort 2: Objective response rate (ORR) per RECIST 1.1 assessed by BICR | Up to approximately 6 years
  The time from randomization to date of first documentation of disease progression or death.

SECONDARY OUTCOMES:
Cohort 1: ORR per RECIST 1.1 assessed by BICR | Up to approximately 6 years
  The time from randomization to date of first documentation of disease progression or death.
Cohorts 1 and 2: ORR per RECIST 1.1 assessed by Investigator | Up to approximately 6 years
  The time from randomization to date of first documentation of disease progression or death.
Cohorts 1 and 2: Overall survival (OS) rate | Up to approximately 7 years
  The time from randomization to date of death from any cause.
Cohorts 1 and 2: Duration of response (DoR) per RECIST 1.1 assessed by BICR | Up to approximately 6 years
  The time from time of first documentation of objective response that is subsequently confirmed to date of first documentation of objective tumor progression or death.
Cohorts 1 and 2: DoR per RECIST 1.1 assessed by Investigator | Up to approximately 6 years
  The time from time of first documentation of objective response that is subsequently confirmed to date of first documentation of objective tumor progression or death.
Cohorts 1 and 2: Disease control rate (DCR) per RECIST 1.1 assessed by BICR | Up to approximately 6 years
  The time from randomization to date of first documentation of disease progression or death.
Cohorts 1 and 2: DCR per RECIST 1.1 assessed by Investigator | Up to approximately 6 years
  The time from Cycle 1 Day 1 to date of first documentation of disease progression or death
Cohorts 1 and 2: PFS per RECIST v1.1 assessed by Investigator | Up to approximately 6 years
  The time from randomization to date of first documentation of disease progression or death.
Cohort 2: PFS per RECIST v1.1 assessed by BICR | Up to approximately 6 years
  The time from randomization to date of first documentation of disease progression or death.
Cohorts 1 and 2: Number of participants reporting adverse events (AEs) and Serious adverse events (SAEs) | Until 30 days post last dose, up to approximately 6 years
Cohorts 1 and 2: Number of Participants with Clinically Significant Changes in Laboratory Results | Until the end of treatment, up to approximately 6 years
Cohorts 1 and 2: Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) | Until the end of treatment, up to approximately 6 years
Cohorts 1 and 2: Number of Participants with Clinically Significant Changes in vital signs | Until the end of treatment, up to approximately 6 years
Cohorts 1 and 2: Change from Baseline in Euroqol-5 Dimensions (EQ-5D) Questionnaire | Until the end of treatment, up to approximately 6 years
Cohorts 1 and 2: Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Until the end of treatment, up to approximately 6 years

CONTACTS AND LOCATIONS:
Locations (170):
- United States (32):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Virginia K. Crosson Cancer Center at St. Jude Medical Center, Fullerton, California
  - University of California - Irvine Medical Center, Orange, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Adventist Health St. Helena, St. Helena, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - AP Medical Research, Miami, Florida
  - Mount Sinai Medical Center of Florida, Inc., Miami Beach, Florida
  - Moffitt, Tampa, Florida
  - Southern Illinois University (SIU) - Simmons Cancer Institute, Springfield, Illinois
  - Mission Cancer + Blood, Des Moines, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - UofL Health Brown Cancer Center, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Corewell Health, Grand Rapids, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - XCancer Omaha/Urology Cancer Center, Omaha, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - Summit Health (New Jersey Urology), Voorhees Township, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical University of South Carolina (MUSC) - Hollings Cancer Center, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Argentina (10):
  - Centro de Diagnostico Urologico S.R.L., Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital Sirio Libanes de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Fundacion Medica Rio Negro y Neuquen, Cipolletti
  - Centro Medico Privado (CEMAIC), Córdoba
  - Fundación CORI para la investigación y Prevención del Cancer, La Rioja
  - Centro De Investigacion Pergamino S.A., Pergamino
  - Instituto de Oncologia de Rosario, Santa Fe
  - Clinica Viedma S.A., Viedma
- Australia (11):
  - Cancer Research SA, Adelaide
  - Mater Misericordiae Ltd, South Brisbane, Brisbane
  - Townsville Hospital and Health Service, Douglas
  - Barwon Health, Geelong
  - Calvary Mater Newcastle, Hunter
  - Sir Charles Gairdner Hospital, Nedlands
  - Blacktown Hospital, New South Wales
  - Prince of Wales Hospital, Randwick
  - Icon Cancer Centre, South Brisbane
  - Gold Coast University Hospital, Southport
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Urologie und Andrologie Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Krankenhaus der Barmherzigen Brüder Wien, Vienna
  - Medizinische Universitaet Wien, Vienna
- Belgium (4):
  - ASBL Grand Hôpital de Charleroi (GHdC), Site Notre Dame, Charleroi
  - General Hospital Maria Middelares, Ghent
  - University Hospital Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (7):
  - Fundacao PIO XII - Hospital de Amor, Barretos
  - CEPEN - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina, Florianópolis
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia, Ijuí
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa, Porto Alegre
  - Hospital Sao Lucas - Pontificia Universidade Catolica do Rio Grande do Sul (PUCRS), Porto Alegre
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital A.C. Camargo Cancer Center, São Paulo
- Canada (4):
  - British Columbia Cancer Agency- Centre for the Southern Interior, Kelowna
  - McGill University Health Center, Québec
  - Princess Margaret Hospital, Toronto
  - Cancer Care Manitoba, Winnipeg
- Chile (3):
  - Fundación Arturo López Pérez (FALP), Santiago
  - Centro de Investigacion Clinica Bradford Hill, Santiago
  - Oncocentro APYS, Viña del Mar
- Aalborg University Hospital, Aalborg, Denmark
- France (15):
  - Service d'Oncologie Medicale - CHRU Besancon, Besançon
  - CHU Bordeaux - Hopital Saint-Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Groupement de Cooperation Sanitaire (GCS) ELSAN - Clinique Victor Hugo, Le Mans
  - CHU de Limoges - Hopital Dupuytren 1, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - ICM - Institut Regional du Cancer de Montpellier, Montpellier
  - Centre d'Oncologie de Gentilly, Nancy
  - Centre Antoine-Lacassagne, Nice
  - Institut Mutualiste Montsouris, Paris
  - AP-HP Hopital Europeen Georges Pompidou, Paris
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers - Pole Regional de Cancerologie de Poitiers (PRC), Poitiers
  - Institut Gustave Roussy, Villejuif
- Georgia (4):
  - LTD High Technology Hospital Medcenter, Batumi
  - The First University Clinic of Tbilisi State Medical University, Tbilisi
  - New Vision University Hospital, Tbilisi
  - Multiprofile Clinic Consilium Medulla LTD, Tbilisi
- Germany (11):
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Universitaetsklinikum Frankfurt - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Georg-August-Universitaet Goettingen Stiftung oeffentlichen Rechts Universitaetsmedizin Goettingen, Göttingen
  - Marien Hospital Herne - Universitaetsklinikum der Ruhr-Universitaet Bochum, Herne
  - Universitaetsmedizin Mannheim, Mannheim
  - Universitaetsklinikum Muenster, Münster
  - Studienpraxis Urologie, Nürtingen
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (4):
  - Orszagos Onkologiai Intezet, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét
- Israel (6):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Rambam Health Care Campus, Haifa
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Centro Riferimento Oncologico - Aviano, Aviano
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Poland (4):
  - Copernicus PL Sp. z o.o., Wojewodzkie Centrum Onkologii, Gdansk
  - Spitale Pomorskie Sp.z.o.o ODDZIAL ONKOLOGII KLINICZNEJ, Gdynia
  - SCM Sp. z o.o., Krakow
  - Mazowiecki Szpital Onkologiczny, Wieliszew
- University Clinical Center of Serbia, Clinic of Urology, Belgrade, Serbia
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (8):
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang
  - Chonnam National University Hwasun Hospital, Gwangju
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (14):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Instituto Valenciano de Oncologia, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital (CGMHLK), Taoyuan
- Turkey (Türkiye) (6):
  - Liv Hospital Ankara, Ankara
  - Trakya University Medical Faculty, Edirne
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Istinye Universitesi VM Medical Park Pendik Hastanesi, Istanbul
  - Medical Point Izmir Hospital, Izmir
  - Kocaeli University Faculty of Medicine, Kocaeli
- United Kingdom (9):
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - St. Bartholomew's Hospital, London
  - University College London Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Derriford Hospital, Plymouth
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No